CLINICAL TRIAL: NCT02795130
Title: Short-Term Outcomes of Different Suture Materials for Sclerotomy Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160382
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Ophthalmologic Surgical Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8-0 polyglactin 910 (Experimental)
  Interventions: Procedure: Sclerotomy closure
- 6-0 plain gut suture (Experimental)
  Interventions: Procedure: Sclerotomy closure

INTERVENTIONS:
Procedure: Sclerotomy closure — Comparison between two suture materials: 1) 8-0 polyglactin 910, 2) 6-0 plain gut

SUMMARY:
Small-incision vitrectomy techniques have become increasingly popular, with a number of advantages over the older 20-gauge instrumentation. The beveled wounds created by the 23- and 25-gauge trocar systems theoretically do not require sutured closure. However, a certain fraction of cases, 1% for 25-gauge systems, and 4-38% for 23-gauge systems, do require suture placement. Poor wound closure puts the patient at increased risk of post-operative hypotony and is associated with increased risk of endophthalmitis. Currently, surgeons are divided as to which suture is the best for sclerotomy closure. The current standard of care is 8-0 polyglactin 910 (Vicryl, Ethicon, Cincinnati, OH). This suture is soft and easy to work with; however, it triggers a robust inflammatory response. The alternative is 6-0 plain gut suture, which is more difficult to manipulate and thicker, but causes less tissue inflammation1. The purpose of this study is to prospectively evaluate these two options for sclerotomy closure. The results of this study will enable us to minimize patients' post-operative discomfort while maximizing safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Dr. Michael Dollin
* Age 18 years and older
* Scheduled to undergo 23-gauge pars plana vitrectomy for any indication that would most likely require sutures (E.g. retinal detachment)

Exclusion Criteria:

1. History of previous vitrectomy in the study eye
2. History of scleral buckling in the study eye
3. Currently on peri-operative corticosteroid medicines (topical or systemic)
4. Systemic chemotherapy within the preceding 6 months.
5. History of any disorder or medication use associated with conjunctival, scleral, or episcleral inflammation and/or scarring
6. History of narcotic abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Patient comfort | 1 month
  One month post-operative patient comfort assessed using a 0-10 visual analogue scale

SECONDARY OUTCOMES:
Scleral/conjunctival inflammation | 1 month
  Rated on a 0 to 4+ scale
Visual Acuity | 1 month
Intraocular Pressure | 1 month
Complications | 1 month

IPD SHARING:
Plan to Share IPD: Yes